CLINICAL TRIAL: NCT04489966
Title: Effects of Aerobic Training on Pancreatic Fat and Cognitive Function in Patients With Type 2 Diabetes
Brief Title: Effects of Aerobic Training on Pancreatic Fat and Cognitive Function in T2DM Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Lou Qingqing, Director of Health Education Department, Nanjing University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019LWKY009
Record Dates: First submitted 2020-07-17; First posted 2020-07-28 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: aerobic training; type 2 diabetes mellitus; pancreatic fat content; cognitive function; hippocampal volume
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Aerobic training group (Experimental): The aerobic training group was performed 3 times/week for 60 minutes/session(including 5 minutes of warm-up, 50 minutes aerobic rhythmic exercise and 5 minutes to relax) for moderate(60 to 70% of participants' HRmax) aerobic rhythmic exercise. All patients received an open class, relate to diabetes health education. The intervention lasted for 6 months.
  Interventions: Behavioral: Aerobic training
- Control group (No Intervention): Patients in control group remained the original lifestyle unchanged. All patients received an open class, relate to diabetes health education.
- Intervention group (Experimental): The intervention was aerobic rhythmic exercise, with intensive training under the guidance and supervision of a professional.The aerobic training program required participants to exercise 3 days/week for 60 minutes/session (including 5-10 minutes of warm-up and 5-10 minutes flexibility exercises). Participants were educated on aerobic exercises (aerobic dancing) with music.The intervention lasted for one year.
  Interventions: Behavioral: Aerobic training
- Compared group (No Intervention): The control group was instructed to maintain their usual habits and received no structured exercise intervention. But the form, frequency and time of movement of each participant must be recorded.Participants receive an open diabetes health education class once a month, which is taught by a specially trained diabetes nurse.

INTERVENTIONS:
Behavioral: Aerobic training — The intervention was aerobic rhythmic training under the guidance and supervision of a professional. The aerobic training program required participants to exercise 3 days/week for 60 minutes/session (including 5-10 minutes of warm-up and 50 minutes aerobic training and 5-10 minutes to relax). All patients received an open class, relate to diabetes health education．
  Arms: Aerobic training group; Intervention group

SUMMARY:
The primary aim of this study was to evaluate the difference in cognitive function and brain functional structure between exercise group and control group by performing regular one-year moderate-intensity aerobic training in type 2 diabetes mellitus (T2DM) with normal cognitive function. The secondary aim of this study was to explore the effects of six-month regular moderate-intensity aerobic training on pancreatic fat content, metabolic index of glucose and lipid, as well as cardiovascular risks in patients type 2 diabetes mellitus.

DETAILED DESCRIPTION:
In recent years, more attention has been paid to the role of aerobic exercise in improving cognitive ability, but there is still a lack of prospective studies on the T2DM population with normal cognitive function. Therefore, the purpose of this study is to compare the differences of cognitive function and hippocampal volume between exercise group and non-exercise group by regular moderate-intensity aerobic exercise intervention for one year in T2DM patients with normal cognitive function to evaluate the impact of aerobic exercise on cognitive function and hippocampal volume for these patients and provide scientific evidence for early prevention and delaying the occurrence of cognitive dysfunction in patients with T2DM. Pancreatic fat deposition in patients with type 2 diabetes is not only a simple fat accumulation but also an early marker of insulin resistance. In this study, The effectiveness of six months of an aerobic exercise intervention on pancreas fat reduction for type 2 diabetes patients was examed.

In this study, 106 T2DM patients who met the inclusion criteria were enrolled and randomized into two groups. All patients received diabetes education(once a month, the course will be focused on basic knowledge of diabetes, diet management, and blood glucose monitoring). The control group followed their regular lifestyle without exercise intervention and recorded 24-hour dietary intake. The aerobic training group was supervised by the trainers who had received professional training and given 60min moderate aerobic rhythmic exercise (including 5min warm-up, 50min aerobic exercise, and 5min stretching exercise).

Baseline assessment included demographic data, duration of diabetes, body mass index（BMI）, waist circumference（WC）, hip circumference（HC）, systolic blood press（SBP）, diastolic blood press（DBP）, smoking and drinking, drug use, acute and chronic complications of diabetes, other chronic complications, 24-hour diet review, international physical activity questionnaire (IPAQ).

Evaluation after 6 months of intervention included pancreatic fat content(PFC), liver fat content (LFC), visceral adipose tissue (VAT), subcutaneous adipose tissue(SAT), fasting plasma glucose (FPG), 2-hour postprandial blood glucose(2hPG), hemoglobin A1c(HbA1c), fasting insulin (FINS), homeostasis model assessment of insulin resistance(HOMA2-IR), homeostasis model assessment of Beta-cell function (HOMA2-β), early insulin secretion index(Δ I30 / Δ G30), total cholesterol(TC), triglycerides(TG),high-density-lipoprotein-cholesterol(HDL-C),low-density lipoprotein cholesterol(LDL-C). The Framingham cardiovascular risk scale (Framingham) and 10-year ischemic cardiovascular disease risk assessment (ICVD) scores were calculated.

Evaluation after 12 months of intervention included fasting plasma glucose(FPG),30 minutes postprandial glucose(30minPG), 2-hour postprandial glucose(2hPG)，hemoglobin A1c(HbA1c), fasting insulin(FINS),30 minutes Insulin(30minINS), homeostasis model assessment of insulin resistance(HOMA2-IR),homeostasis model assessment of Beta cell function(HOMA2-β),early insulin secretion index(Δ I30 / Δ G30),totalcholesterol(TC),triglycerides(TG),high-density-lipoprotein cholesterol( HDL-c），low-density-lipoprotein cholesterol(LDL-c),muscle mass, right, left hippocampal volume of hippocampal volume, the hippocampal volume, and total physical activity energy expenditure, total moderate physical activity energy expenditure. In addition to this, cognitive function (MMSE, MoCA) were also evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed of T2DM based on the 1999 diagnostic criteria of the WHO;
2. Had normal muscle strength; 3.18.5≤BMI≤35kg/m2;

4.Had normal cognitive function ( MMSE ≥27 points, MoCA ≥26 points) ; 5.Primary school education or above ( Participants were able to fill in the scale) ; 6.Aged 60-75 years; 7.Had ≥5 years duration of T2DM; 8.Had no evidence of hearing or visual impairment and communication difficulties; 9.Were willing to participate in the study and signed informed consent voluntarily.

Exclusion Criteria:

1. With severe acute complications of diabetes;
2. Serious heart, liver and kidney dysfunction, and cardiovascular and cerebrovascular diseases, such as cerebral infarction, cerebral hemorrhage, etc.;
3. Pregnant and lactating women;
4. Sleep disorders (PSQI >7 points);
5. Had a family history of dementia;
6. Alcohol dependence and oral medications that affect cognitive function (such as antipsychotic drugs, sedative hypnotics, etc.);
7. Contraindications for MRI, such as metal implant in the body.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
Cognitive function scale(1) | 12 months
  Mini-mental State Examination(MMSE) includes five aspects: orientation, memory, attention and calculation, recall and language ability, with a total score of 30.The scoring standard is: 27-30 is normal;< 27 was divided into cognitive impairment;Mild cognitive impairment ≥21 and < 27 points;Moderate cognitive impairment 10-20;Severe cognitive impairment ≤9, the higher the score, the better the cognitive function.
Cognitive function scale(2) | 12 months
  The Montreal Cognitive Assessment Scale (MoCA) includes eight aspects: visuospatial and executive function, nomenclature, memory, attention, language, abstraction, delayed recall, and orientation for a total of 30 points.The score criteria are as follows: ≥26 is considered as normal cognitive function; < 26 is considered as cognitive dysfunction. If the number of years of education ≤12 years, the score is added 1 point to correct cultural influence. The lower the score, the worse the cognitive function.
Brain functional structure---Hippocampal volume | 12 months
  Hippocampal volume measurement by the same operation, all patients using 3D brain volume sequence (3D - BRAVO) image data acquisition of high resolution T1W1 brain structure, specific scanning parameters is as follows: repetition time (TR) = 9.5 ms, Time of Echo(TE) = 3.9 ms, Flip angle (FA) = 12 °, matrix=320 x 320, scanned area (FOV) = 22 x 22 cm, depth of stratum=1.5mm, interlamellar spacing =1.5mm.
Abdominal fat Abdominal fat | 6 months
  Pancreatic fat content（PFC,%）

SECONDARY OUTCOMES:
Glycemic control(1) | 12 months
  Fasting Plasma Glucose(FPG, mmol/L)
Glycemic control(2) | Time Frame: 12 months
  2-hour postprandial blood glucose (2hPG, mmol/L)
Hemoglobin A1c | 12 months
  Hemoglobin A1c(HbA1c,mml/ml)
HOMA2-IR and HOMA2-β | 12 months
  Homa-IR is an indicator used to assess an individual's level of insulin resistance, HOMA-β is used to evaluate the function of individual islet cells, ΔI30/ΔG30（The ratio of net insulin to glucose increment 30 min after glucose load）
Blood lipids | 12 months
  Total Cholesterol(TC,mmol/L),Triglycerides(TG,mmol/L), High-density-lipoprotein Cholesterol(HDL-c,mmol/L), Low-density-lipoprotein Cholesterol(LDL-c,mmol/L)
Other abdominal fat(1) | 6 months
  Liver fat content(LFC,%)
Other abdominal fat(2) | 6 months
  Visceral adipose tissue(VAT,cm²)
Other abdominal fat(3) | 6 months
  Subcutaneous adipose tissue(SAT,cm²)
The international physical activity questionnaire | 6 months
  The international physical activity questionnaire (IPAQ) content mainly includes five aspects: physical activity of the relevant related work (including high levels of physical activity, moderate physical activity, walking), traffic-related physical activity (including bus, ride a bike, on foot), housework on physical activity (courtyard in heavy physical activity, physical activity among the courtyard, indoor physical activity), entertainment and leisure-time physical activity (walking, heavy physical activity, moderate physical activity) and meditation time. Participants were asked to recall the amount of time spent in each type of activity during the past week, including the number of days during the week and the number of hours spent each day, and to assign MET values to each type of physical activity using the MTE table. Energy consumption (MEt-min /week) for each type of physical activity = metabolic value of the activity (MET) × activity time per day (min) × activity days /week
The Framingham Cardiovascular Risk Scale | 6 months
  The Framingham Cardiovascular Risk Scale is used to predict 10-year cardiovascular disease severity, cardiovascular event risk, and risk stratification. The scale includes 6 risk factors, including gender, age, TC, HDL-C, SBP, and smoking status. The total score was determined according to gender, then the corresponding scores were determined according to age, TC, HDL-C, SBP, and smoking status. The total score was calculated by adding up, and then the 10-year incidence risk of CHD corresponding to the total score was looked up. 10-year cardiovascular risk of < 10% is a low risk, 10-20% is a moderate risk, and > 20% is a high risk.
The 10-year risk assessment table for Ischemic cardiovascular disease | 6 months
  The 10-year risk assessment table for Ischemic cardiovascular disease (ICVD) in Chinese people was used to calculate the 10-year risk of ICVD. The scores of men and women were selected based on their gender, and the corresponding scores of age, systolic blood pressure, BMI, TC, smoking, and diabetes were checked in the table. Then the total score was calculated and the absolute risk of ICVD was checked according to the total score (%). The 10-year risk of ICVD is very low, 5%-10% is low, 10%-20 is moderate, 20%-40% is high, and ≥40% is very high.

CONTACTS AND LOCATIONS:
Overall Officials: Qingqing Lou, PhD, Principal Investigator — Nanjing University of Traditional Chinese Medicine
Locations (1):
- Affiliated Hospital of Integrated Traditional Chinese and Western Medicine, Nanjing University of Chinese Medicine, Nanjing, Jiangsu, China

REFERENCES:
- [Result] Alberti KG, Zimmet PZ. Definition, diagnosis and classification of diabetes mellitus and its complications. Part 1: diagnosis and classification of diabetes mellitus provisional report of a WHO consultation. Diabet Med. 1998 Jul;15(7):539-53. doi: 10.1002/(SICI)1096-9136(199807)15:73.0.CO;2-S. PMID 9686693
- [Derived] Wang Y, Wang L, Yan J, Yuan X, Lou QQ. Aerobic Training Increases Hippocampal Volume and Protects Cognitive Function for Type 2 Diabetes Patients with Normal Cognition. Exp Clin Endocrinol Diabetes. 2023 Nov;131(11):605-614. doi: 10.1055/a-2105-0799. Epub 2023 Jun 2. PMID 37268011